CLINICAL TRIAL: NCT07021417
Title: Effectiveness of Primary Care Nurse-supervised Educational Group Interventions for Giving up Smoking: A Randomized Con-trolled Trial
Brief Title: Effectiveness of Primary Care Nurse-supervised Educational Group Interventions for Giving up Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 06052025; FFIS17/CE/01/26 (Other Grant/Funding Number: Fundación Formación-Investigación Sanitaria of Murcia)
Record Dates: First submitted 2025-05-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Smoking Cessation
Keywords: Nurses; Nursing Evaluation Research; Primary Health Care; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop (Experimental): Format:
  A single group session of four hours' duration.
  Structure:
  All content and activities were concentrated into a single meeting.
  Methodology:
  Cognitive-behavioural techniques and participatory dynamics were employed, fostering motivation and vicarious learning among group members.
  Focus:
  The initial parts of the session were oriented towards preparing participants for smoking cessation, whilst the final segment focused on maintaining abstinence and preventing relapse.
  Materials:
  A standardised presentation and a procedural guide were utilised to ensure the homogeneity of the intervention.
  Digital Support:
  All participants received instructions on how to use the S'Acabó mobile application as a complement to the workshop.
  Interventions: Behavioral: Workshop
- Course (Experimental): Format:
  A group programme comprising four weekly sessions of two hours each (eight hours in total).
  Structure:
  Sessions were distributed over the course of one month, allowing for a more gradual and sustained accompaniment.
  Methodology:
  Cognitive-behavioural techniques and participatory strategies were applied, facilitating the exchange of experiences and mutual support among participants.
  Focus:
  The first two sessions focused on preparation for smoking cessation, while the third and fourth sessions were dedicated to maintaining abstinence and preventing relapse.
  Materials:
  The same standardised materials and procedural guides as those used in the single workshop were employed.
  Digital Support:
  Use of the S'Acabó mobile application was also recommended as reinforcement for the content addressed in the face-to-face sessions.
  Interventions: Behavioral: Course

INTERVENTIONS:
Behavioral: Workshop — includes a single 4-hour session
  Arms: Workshop
Behavioral: Course — Includes four weekly sessions totaling 8 hours (2 hours each)
  Arms: Course

SUMMARY:
Background: To analyze the effectiveness of two group interventions for smoking cessa-tion (with support from the app) conducted by primary care nurses. Methods: A multi-center randomized controlled clinical trial occurred across eight Health Centres in the Murcia Region from 2018 to 2019. It involved daily smokers aged 18 and older who wanted to quit, had internet access, and spoke Spanish. Pregnant women, polydrug users, and individuals with psychiatric disorders were excluded from participation. Participants were randomly divided into two groups: one attending a single 4-hour Workshop, and the other attending a Course consisting of four 2-hour sessions. The analysis of smoking abstinence was performed using SPSS V22, with intragroup differences assessed through the chi-square test.

DETAILED DESCRIPTION:
The project was conceived as a randomised, multicentre clinical trial aimed at comparing the efficacy of two group-based intervention modalities for smoking cessation, both led by primary care nurses and supplemented by using the S'Acabó mobile application. The study was conducted in health centres across the Region of Murcia between 2018 and 2019, with participants being followed up for one year. The target population comprised adult smokers who expressed a desire to quit smoking, had internet access, and did not present with severe psychiatric disorders or concurrent substance use.

Allocation to the intervention groups was performed randomly: one group participated in a single four-hour workshop, whilst the other attended a course consisting of four weekly sessions, each lasting two hours. Both modalities incorporated cognitive-behavioural techniques and participatory methodologies to enhance individual motivation and group learning through the exchange of experiences and peer support.

The nurses responsible for delivering the interventions received specific training in smoking cessation, group education, and the management of group dynamics, thereby ensuring the standardisation and quality of the process. The study protocol included the systematic collection of sociodemographic, clinical, and tobacco consumption data, the assessment of psychological variables and the utilisation of complementary resources, including the mobile application. Follow-up of participants was conducted through face-to-face visits and telephone contacts at various points throughout the year, enabling the monitoring of the smoking cessation process and adherence to the proposed strategies. Statistical analysis of the data was carried out by international methodological standards, employing validated tools and ensuring the robustness and reliability of the results obtained.

ELIGIBILITY:
Inclusion criteria:

* Daily smokers aged over 18 years.
* Smoking history of at least one year.
* Intention to quit smoking within one month.
* Ability to communicate in Spanish.
* Ownership of a mobile device with internet access.

Exclusion criteria:

* Consumption of other drugs (excluding cannabis).
* Participation in smoking cessation programmes within the past year.
* Diagnosis of an acute psychotic disorder.
* Adolescents.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who are abstinent (self-reported abstinence corroborated by an exhaled carbon-monoxide reading, expressed in parts per million). | Up to 12 months post-intervention (telephone contacts at months 3 and 9; face-to-face visits with carbon-monoxide testing at months 6 and 12).
  Assessment of effectiveness: Abstinence rates for the Course and the Workshop groups will be compared by means of the χ² test at 3-, 6-, 9- and 12-month follow-ups. Data will be analysed with SPSS v22; statistical significance will be set at p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida Lozano-Polo, Phd, Principal Investigator — Universidad de Murcia
Locations (1):
- Faculty of Nursing, Cartagena, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT07021417/Prot_000.pdf